CLINICAL TRIAL: NCT05604222
Title: Effect of Behavioral Sleep Intervention on Lower Urinary Tract Symptoms in Older Women
Acronym: SLAB
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shachi Tyagi (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Shachi Tyagi, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY22050099; 1R01AG076575-01 (NIH)
Record Dates: First submitted 2022-10-12; First posted 2022-11-03 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Urgency Urinary Incontinence; Nocturia
MeSH Terms: conditions — Nocturia | interventions — mirabegron

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirabegron (Experimental): Mirabegron for 8 weeks
  Interventions: Drug: Mirabegron 50 MG
- Mirabegron plus Brief Behavioral Treatment for Insomnia (BBTI) (Experimental): Mirabegron for 8 weeks and a 4 week behavioral intervention for insomnia
  Interventions: Drug: Mirabegron 50 MG; Behavioral: Brief Behavioral Treatment for Insomnia

INTERVENTIONS:
Drug: Mirabegron 50 MG — Medication to treat overactive bladder
  Other Names: Myrbetriq
Behavioral: Brief Behavioral Treatment for Insomnia — A behavioral intervention for insomnia
  Other Names: BBTI
  Arms: Mirabegron plus Brief Behavioral Treatment for Insomnia (BBTI)

SUMMARY:
Urgency urinary incontinence (UUI) is common in older people and vastly reduces quality of life, yet the cause and mechanism of disease are not well understood. This study will investigate the role of adding behavioral sleep intervention to the standard pharmacotherapy in treatment of UUI among older adults, and the brain mechanisms involved in continence by evaluating brain changes. This will expand the current knowledge of how the sleep affects bladder control, and better characterize the brain mechanisms in maintaining continence.

DETAILED DESCRIPTION:
Urgency urinary incontinence (UUI), a form of overactive bladder (OAB), is prevalent (36% of women over age 65), morbid and costly ($83 billion/year), and treatment is problematic. Current treatment is largely bladder centric has limited efficacy,and adherence rates fade to 21% at 12 months. The researchers believe that a complimentary approach, one that also addresses etiology beyond the bladder may enhance treatment success. Up to 50% of older adults complain of poor sleep and nighttime bladder symptoms (nocturia) are considered the major cause. However, the relationship between sleep and the bladder is complex and bidirectional. Poor sleep not only exacerbates daytime lower urinary tract symptoms (LUTS), but can also cause these, increasing the risk of LUTS by up to 55% over 5 years. Sleep disruption increases anxiety and impairs daytime attention, both of which affect bladder control. Consistent with findings in anxiety disorders and attention control, poor sleep is linked to media prefrontal cortex (mPFC) hypoactivity, a region the investigators have identified as key to executive control of voiding and to therapeutic response to biofeedback-assisted pelvic floor muscle therapy. Hence, the investigators posit that enhanced mPFC function through improved sleep might ameliorate bladder control. Despite evidence of a bidirectional relationship, the impact of sleep treatment on UUI has never been assessed. The researchers prior study demonstrated that improving sleep using Brief Behavioral Treatment of Insomnia (BBTI), a simple intervention for insomnia, improved both sleep and nocturia in older adults, yet its impact on UUI and mechanism of action is not known. Our exploratory analysis of sleep and voiding data from 20 older adults with UUI and nocturia showed that with behavioral sleep intervention alone, 24-hour UUI episodes decreased with prolongation of uninterrupted sleep before the first awakening to void (r=-0.50, p=0.02), and increased proportion of deep sleep (r=-0.56, p=0.01). Hence, the researchers postulate that addressing sleep in patients with UUI and nocturia may further potentiate bladder-focused UUI treatment. The efficacy of mirabegron, a β3- adrenoceptor agonist is comparable to first-line antimuscarinic pharmacotherapy for UUI, with fewer side effects, but it has only a modest effect on nocturia. Although these drugs show statistically significant improvement in LUTS, drug compliance remains poor secondary to modest perceived clinical benefit. The researchers central hypothesis is that comorbid insomnia contributes to poor therapeutic response for UUI and concurrent insomnia treatment will improve outcomes. Specifically, addition of BBTI to drug therapy will improve sleep, nocturia, and daytime LUTS, likely mediated by improvement of mPFC function.

The researchers propose an 8-week randomized controlled trial of mirabegron+BBTI vs. mirabegron alone for UUI in 100 women (aged ≥60), assessing both clinical and neural effects of treatment. The researchers will also assess durability of the combination therapy at 6 months. This design encompasses the role of sleep in OAB treatment, insight into the central and peripheral effects of mirabegron and BBTI, and response durability.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory women aged 60+ years
* urgency incontinence or urge-predominant mixed incontinence (able to differentiate between stress symptoms-cough, laugh, exercise-and leakage following the sudden onset of a strong urge to void that is difficult to defer during questioning on telephone screening) occurring at least five times weekly for ≥ 3 months despite treatment for reversible causes
* nocturia ≥2 each night
* subjects with current or previous use of anticholinergic medications will be considered for the study if willing to go through a washout period of at least 4 weeks of duration

Exclusion Criteria:

* contraindication to any of the drugs used (e.g., mirabegron, prophylactic antibiotics)
* cognitive impairment (MOCA score <24 or inability to accurately complete a voiding diary, perform a 24-hour pad test, reliably take daily medication, or comply with fMRI testing)
* prior treatment with intradetrusor onabotulinum toxin or sacral neuromodulation.
* spinal cord injury; history of pelvic irradiation, advanced uterine or bladder cancer; multiple sclerosis
* urethral obstruction; urinary retention [PVR >200 ml]
* interstitial cystitis; artificial sphincter implant
* medical instability or expected change in medication during the study
* conditions that preclude fMRI testing, such as history of claustrophobia, history or suspicion of implanted metal or electronic object
* requirement for intravenous antibiotics for bacterial endocarditis prophylaxis or presence of multiple allergies to the antibiotics available in our protocol
* chronic or recurrent bowel issues, e.g. IBS, colitis, fecal incontinence
* known allergy to study medication or interaction with current medications
* severe uncontrolled hypertension >180 mmHg systolic or >100 mmHg diastolic

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Potential participants must be biologically female
Enrollment: 120 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Incontinence episodes | Baseline to 8 weeks
  The number of incontinence episodes

SECONDARY OUTCOMES:
Structural brain changes | Baseline to 8 weeks
  Change in grey and white matter volume on MRI compared between the two arms. Grey matter and white matter volume of important brain structures will be compared via tractography.
Functional brain changes | Baseline to 8 weeks
  Change in brain functional response to an infusion/withdrawal protocol compared between the two arms. Changes are displayed as a map of t-values for each voxel of the brain, showing likelihood of statistical significance of changes.
Nocturia episodes | Baseline to 8 weeks
  The number of nocturia episodes

CONTACTS AND LOCATIONS:
Overall Officials: Shachi Tyagi, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification may be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following publication, no end date
Access Criteria: Any purpose